CLINICAL TRIAL: NCT01841021
Title: Pilot Study of Brentuximab Vedotin in Relapsed/Refractory Peripheral T-Cell Lymphoma Expressing CD30 Receptor
Brief Title: Pilot Study of Brentuximab Vedotin in Relapsed/Refractory Peripheral T-Cell Lymphoma Expressing CD30
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual, loss of sponsor support
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17343; 35-IST-019 (Other Grant/Funding Number: Seattle Genetics)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Peripheral T-Cell Lymphoma (PTCL); Relapsed; Refractory; CD30 Receptor; Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence | interventions — Brentuximab Vedotin; Immunoconjugates; Drug Therapy; monomethyl auristatin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin Treatment (Experimental): Brentuximab vedotin will be given intravenously with a dose of 1.8 mg/kg every 21 days, over 30 minutes for 16 cycles in the clinic.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin will be given by intravenous infusion (into a vein) on Day 1 of every 21 day cycle.
  Other Names: SGN-35; ADCETRISTM; antibody drug conjugate(ADC); chemotherapy; monomethyl auristatin E (MMAE)

SUMMARY:
The main purpose of this study is to test if brentuximab vedotin has an effect on cancer in patients with a certain type of large B-cell lymphoma. The side effects (unwanted effects) of SGN-35 in patients with this certain type of large B-cell lymphoma will also be studied. It is not known if brentuximab vedotin is better or worse than other treatment patients might be given.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PTCL expressing CD30 receptor. Following PTCL subtypes will be eligible: Peripheral T - cell lymphoma, not otherwise specified (NOS); Angioimmunoblastic T-cell Lymphoma; Subcutaneous Panniculitis Like T-cell Lymphoma; Hepatosplenic gamma/delta T cell Lymphoma; Extranodal natural killer (NK)T-cell Lymphoma, nasal type; Enteropathy-associated T-cell lymphoma; Adult T-cell Leukemia/lymphoma; T-cell prolymphocytic leukemia; Primary cutaneous gamma-delta T-cell lymphoma; Aggressive NK cell leukemia; Aggressive subtype of T cell Large Granular Lymphocytic (LGL) or transformed LGL leukemia; Epstein Barr Virus(EBV)-positive T-cell lymphoproliferative disorders of childhood; Transformed mycosis fungoides who have progressed following treatment with at least one systemic therapy; Sezary syndrome
* Histology slides and pathology material must be available at the site for each patient before enrollment in order to be sent to the Leading Institution of the study for central pathology review and pharmacodynamic studies.
* Patients must have progressive, relapsed or refractory disease after: At least one prior systemic anti-lymphoma regimen (chemotherapy or immunotherapy except for transformed mycosis fungoides as described previously); Relapsed or failed autologous or allogeneic stem cell transplant.
* Understand and voluntarily sign an Institutional Review Board (IRB) approved informed consent form
* Must have at least one site of disease (index lesion) measurable in two dimensions by computed tomography (CT)
* Patients with leukemic form of PTCL who will not have a measurable lesion in two dimensions by CT scan, relapsed or refractory disease must be detected by immunohistochemistry or flow cytometry and molecular clonality studies in bone marrow or peripheral blood.
* At least 2 weeks since the last chemotherapy, radiation therapy, immunotherapy or any investigational products
* Must meet the following criteria within 4 days before the first dose of study drug:

  * Neutrophils ≥1,000/ul
  * Hemoglobin ≥ 8 g/dL
  * Platelets≥ 50.0x10^9 /L
  * Total bilirubin ≤ 1.5 x upper normal limit, or ≤ 5 x upper normal limit if documented hepatic involvement with lymphoma or history of Gilbert's Syndrome
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper normal limit (≤ 5 x upper normal limit if documented hepatic involvement with lymphoma)
  * Calculated creatinine clearance ≥ 40 mL/min/1.73 m^2 based on Cockcroft and Gault method
  * PT or International Normalization Ratio (INR), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 x upper limit of normal unless patient is receiving anticoagulants. If patient is on anticoagulation therapy, levels should be within therapeutic range.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
  * Negative pregnancy test for women of childbearing potential
  * Recovered (≤ Grade 1 toxicity) from the reversible effects of prior antineoplastic therapy

Exclusion Criteria:

* Any of the following cardiovascular conditions or values within 6 months before the first dose of study drug: Myocardial infarction and the New York Heart Association (NYHA) Class III or IV heart failure
* History of another primary malignancy not in clinical remission; except adequately treated patients with completely resected in situ carcinoma, such as nonmelanoma skin cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear, or localized prostate cancer with prostate-specific antigen (PSA) <1 ng/ml
* Known active cerebral/meningeal involvement with lymphoma. Asymptomatic patients with previously treated and resolved central nervous system (CNS) lymphoma involvement are permitted.
* Prior administration of Brentuximab vedotin
* Corticosteroid monotherapy for lymphoma within 1 week of the first dose of study drug
* Any serious underlying medical condition that, in the opinion of the investigator or medical monitor, would impair the ability to receive or tolerate the planned treatment
* Known hypersensitivity to recombinant proteins, or any component contained in the drug formulation
* Female patients who are lactating or have a positive serum pregnancy test during the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Sokol, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was enrolled in June 2015 at Moffitt Cancer Center. Soon after the accrual of this one participant, the sponsor terminated their support of the project.
Period: Overall Study
Arm/Group | Brentuximab Vedotin Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: 68] | 68 [68 to 68]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR: The proportion of patients with complete response (CR) and partial response (PR). Follow-up assessments after cycle 16 to be done every 12 weeks for up to 24 months. Restaging imaging computed tomography (CT) scans to be repeated 12 and 24 months from the beginning of the follow-up period. Objective disease response (CR and PR) defined according to the modified 2007 International Working Group (IWG) response criteria for non-Hodgkin lymphomas (NHL). CR = Disappearance of all evidence of disease; PR = Regression of measurable disease and no new sites.
Time Frame: Up to 24 months post treatment
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 1
Participants
  Participants with Complete Response | 0
  Participants with Partial Response | 0
  Participants with Stable Disease | 1

2. Secondary Outcome: Time to Response (TTR)
Description: Investigators intended to report median time and its 95% confidence interval estimate using the Kaplan-Meier method, for 20 participants. TTR: The time from the start of treatment to the first time when the measurement criteria for CR or PR are met. Participants who did not have a confirmed response to be censored at the date of the last tumor assessment.
Time Frame: Up to 24 months post treatment
Population: Participants with Complete Response or Partial Response.
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR: The number of days between the first tumor response assessment of objective response (complete response and partial response) to the time of the first tumor response assessment of progressive disease (PD) or death if due to disease progression (date of first PD assessment or death due to disease progression-date of first objective response assessment +1).
Time Frame: Up to 24 months post treatment
Population: Participants with Complete Response or Partial Response.
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Disease Progression (TTP)
Description: Investigators intended to report median time and its 95% confidence interval estimate using the Kaplan-Meier method, for 20 participants. Progressive disease (PD) defined according to the modified 2007 International Working Group (IWG) response criteria for non-Hodgkin lymphomas (NHL).
Time Frame: Up to 24 months post treatment
Population: All participants.
Measure: Number; unit: months
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 1
months | 10

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Investigators intended to report median time and its 95% confidence interval estimate using the Kaplan-Meier method, for 20 participants. Stable disease (SD) defined according to the modified 2007 International Working Group (IWG) response criteria for non-Hodgkin lymphomas (NHL).
Time Frame: 24 months post treatment
Population: Participants evaluable at 24 months post treatment.
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Investigators intended to report median time and its 95% confidence interval estimate using the Kaplan-Meier method, for 20 participants. Radiological assessments to be discontinued at the time of tumor progression or initiation of new anticancer therapy, after which survival to be evaluated every 3 months until 2 years from the start of study treatment or until study closure.
Time Frame: 24 months post treatment or until study closure
Population: Participants evaluable at 24 months post treatment or at study closure.
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Study Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) to be summarized by worst NCI NCI Common Terminology Criteria for Adverse Events (CTCAE) grade.
Time Frame: Up to 24 months post treatment
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin Treatment
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Brentuximab Vedotin Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin Treatment (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Infusion related reaction (General disorders) | 1 (4)
Investigations - Other (Investigations) | 1 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (3)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Planned accrual: 20. Sponsor withdrew support soon after one enrollment. Accrual was terminated; analysis unable to be performed. Participant stopped treatment after 14 cycles due to progressive lymphadenopathy; entered another clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes